CLINICAL TRIAL: NCT05290246
Title: TRE in Type 2 Diabetes Mellitus (See Food Study 3)
Brief Title: TRE in Type 2 Diabetes (See Food Study 3)
Acronym: SFS3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2022-30316
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type2Diabetes
Keywords: Type 2 diabetes; diet intervention; intermittent fasting; caloric restriction; time restricted eating
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (Experimental): daily 8 hour eating window
  Interventions: Behavioral: Time restricted eating
- Caloric Restriction (Active Comparator): reduction of caloric intake by 15%
  Interventions: Behavioral: Caloric reduction

INTERVENTIONS:
Behavioral: Time restricted eating — Limiting daily eating time to an 8 hour window
  Arms: Time restricted eating
Behavioral: Caloric reduction — Cut caloric intake by 15%
  Arms: Caloric Restriction

SUMMARY:
Hyperglycemia in patients with Type 2 Diabetes Mellitus is initially treated with metformin coupled with intentional caloric restriction, which is difficult to sustain due to multiple barriers, including acquiring the necessary knowledge, teaching the intervention, cost of delivery and potential burden on quality of life. In contrast to intentionally restricting calories, time restricted eating (TRE), presents a simplified view of eating focused on restricting the eating window, which allows ad libitum intake per a person's dietary preferences during a daily fixed eating window. This study proposes a 24 week feasibility study to test if TRE is a viable alternative to Caloric Restriction in improving glycemic measures while accounting for weight loss in overweight/obese patients [BMI:25-45 kg/m2] with metformin-only treated Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese adults with metformin-only treated type 2 diabetes
* 18-65 years old
* BMI:25-45 kg/m2
* HbA1c: 6.5-8.5%
* Self-reported weight must be stable [±5 pounds] for at least 3 months prior to the study
* Owns a smartphone.

Exclusion Criteria:

* Active or anticipated pregnancy during the study
* type 2 diabetes treated with medications other than metformin
* presence of eating disorders as noted by screening survey.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in glycemic measures- HbA1c (12w) | 12 weeks
  Change in hemoglobin A1c

SECONDARY OUTCOMES:
Weight change (12w) | 12 weeks
  Change in weight from baseline
Weight change (24w) | 24 weeks
  Change in weight from baseline
Change in glycemic measures- insulin (12w) | 12 weeks
  Change in fasting insulin
Change in glycemic measures- insulin (24w) | 24 weeks
  Change in fasting insulin
Change in glycemic measures- Homeostatic Model Assessment for Insulin Resistance (24w) | 24 weeks
  Change in Homeostatic Model Assessment for Insulin Resistance
Change in glycemic measures- Homeostatic Model Assessment for Insulin Resistance (12w) | 12 weeks
  Change in fasting Homeostatic Model Assessment for Insulin Resistance
Change in glycemic measures- HbA1c (24w) | 24 weeks
  Change in hemoglobin A1c
Change in glycemic measures- glucose (24w) | 24 weeks
  Change in continuous glucose monitoring
Change in glycemic measures- glucose (12w) | 12 weeks
  Change in continuous glucose monitoring
Intervention burden (12w) | 12 weeks
  Participant self-report via survey
Intervention burden (24w) | 24 weeks
  Participant self-report via survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chow, MD, Principal Investigator — University of Minnesota- Division of Endocrinology, Diabetes, and Metabolism
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States